CLINICAL TRIAL: NCT01295437
Title: A Single-surgeon Randomized Study Comparing Three Composite Meshes on Chronic Pain After Lichtenstein Hernia Repair in Local Anesthesia
Brief Title: Comparison of Three Meshes in Lichtenstein Hernia Repair
Acronym: Lichtenstein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Mikkeli Central Hospital (Other)
Responsible Party: Hannu Paajanen, Department of Surgery, Kuopio University Hospital, Kuopio, Finland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lichtenstein hernia repair; Lichtenstein (Other: Etelä-Savon Eettinen tmk ETMK§11)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Pain; Recurrences
Keywords: inguinal hernia, Lichtenstein hernioplasty, chronic pain
MeSH Terms: conditions — Chronic Pain; Recurrence; Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vypro II mesh (Active Comparator): A partly absorbable polypropylene-polyglactin mesh (50g/m2).
  Interventions: Device: Vypro II mesh
- Premilene LP (Active Comparator): A lightweight polypropylene mesh (55 g/m2)
  Interventions: Device: Premilene LP
- Premilene mesh (Placebo Comparator): A conventional polypropylene mesh (82 g/m2)
  Interventions: Device: Premilene mesh

INTERVENTIONS:
Device: Vypro II mesh — partly absorbable mesh
  Other Names: polypropylene-polyglactin mesh
  Arms: Vypro II mesh
Device: Premilene LP — lightweight mesh
  Other Names: lightweight polypropylene
  Arms: Premilene LP
Device: Premilene mesh — A conventional polypropylene mesh (82 g/m2)
  Other Names: polypropylene mesh
  Arms: Premilene mesh

SUMMARY:
Chronic pain may be a long-term problem after inguinal Lichtenstein hernioplasty. The aim of this study was to compare long-term results of hernioplasty using three different meshes (partly absorbable, lightweight polypropylene and thick polypropylene mesh).

DETAILED DESCRIPTION:
Inguinal hernioplasty was performed under local anesthesia in 300 patients in day-case surgery by the same surgeon and exactly by the same surgical technique. The patients were randomized to receive either a partly polypropylene-polyglactin mesh (Vypro II, 100 hernias), a lightweight polypropylene mesh (Premilene LP, 100 hernias) or a conventional densely woven polypropylene mesh (Premilene, 100 hernias). Pain, patients discomfort and recurrences of hernias were carefully followed 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* uni-or bilateral primary or recurrent inguinal hernia
* patients age >18yrs

Exclusion Criteria:

* previous mesh hernioplasty
* femoral hernia
* emergency operation
* allergy to polypropylene

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-03; Primary Completion 2005-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Presence of chronic pain | 5 years
  Pain scores were measured by using a visual analoque scale.

SECONDARY OUTCOMES:
Presence of recurrences | 5 years
  Recurrence of inguinal hernias after Lichtenstein hernioplasty was studies during clinical and ultrasound examination

CONTACTS AND LOCATIONS:
Overall Officials: Hannu EK Paajanen, MD, PhD, Principal Investigator — University Hospital of Kuopio, Finland
Locations (1):
- Hannu Paajanen, Kuopio, Finland

REFERENCES:
- [Background] Paajanen H. A single-surgeon randomized trial comparing three composite meshes on chronic pain after Lichtenstein hernia repair in local anesthesia. Hernia. 2007 Aug;11(4):335-9. doi: 10.1007/s10029-007-0236-1. Epub 2007 May 10. PMID 17492341
- [Derived] Paajanen H, Ronka K, Laurema A. A single-surgeon randomized trial comparing three meshes in lichtenstein hernia repair: 2- and 5-year outcome of recurrences and chronic pain. Int J Surg. 2013;11(1):81-4. doi: 10.1016/j.ijsu.2012.11.020. Epub 2012 Dec 13. PMID 23246868